CLINICAL TRIAL: NCT00932074
Title: A Phase 1/2 Study Evaluating the Safety, Tolerability and Efficacy of KP-413 Topical Ointment in Subjects With Atopic Dermatitis
Brief Title: A Study to Determine the Safety, Tolerability and Efficacy of KP-413 in Subjects With Atopic Dermatitis(AD)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kaken Pharmaceutical (Industry)
Collaborators: Dow Pharmaceutical Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DPSI-KP413-P2-01
Record Dates: First submitted 2009-06-30; First posted 2009-07-02 (Estimated); Last update posted 2012-04-06 (Estimated); Status verified 2012-04

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 3% KP-413 Ointment (Experimental)
  Interventions: Drug: KP-413 Ointment
- 1% KP-413 Ointment (Experimental)
  Interventions: Drug: KP-413 Ointment
- Placebo (Placebo Comparator)
  Interventions: Drug: KP-413 Ointment

INTERVENTIONS:
Drug: KP-413 Ointment — Study drug ointment to be applied topically to the selected treatment areas on the head/neck and torso/limbs twice a day for 4 weeks.

SUMMARY:
The purpose of this study is to assess the safety, tolerability and efficacy of KP-413 topical ointment compared with vehicle ointment in treating adult subjects with atopic dermatitis (AD).

ELIGIBILITY:
Inclusion Criteria:

* Has a clear diagnosis of AD meeting the Hanifin and Rajka criteria for AD that involves both the head/neck and the torso/limbs, and affects 5-30% of the subject's total BSA as determined using the rule of nines
* Has a Baseline IGSS of 3(moderate) or 4(severe) in the selected treatment area on the torso/limbs, and a Baseline IGSS of 2(mild), 3(moderate) or 4(severe) in the selected treatment area on the head/neck.
* Female of childbearing potential has a negative pregnancy test and will be using an effective method of contraception during the study.

Exclusion Criteria:

* Female who is pregnant, nursing an infant, or planning a pregnancy during the study period.
* Has a Baseline oozing/crusting score of 3(moderate) or greater at the selected treatment area on the head/neck or torso/limbs.
* Presence of a concurrent skin condition that could interfere with assessment of treatment.
* Treatment with any investigational drug or device within 30 days or 5 half lives(whichever is longer) prior to the Baseline visit, or concurrent participation in another clinical trial with an investigational drug or device.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2009-07; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Investigator's Global Severity Score(IGSS) | 4 weeks

SECONDARY OUTCOMES:
Plasma levels of KP-413 | 6 weeks
Signs and Symptoms of AD | 4 weeks
Subject's Numerical Rating Scale(NRS) of Pruritus Score | 4 weeks
Percent of AD-affected body surface area (BSA) | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Barry Calvarese, MS, Study Director — Dow Pharmaceutical Sciences
Locations (6):
- United States (6):
  - Michigan Center for Research Corp, Clinton Twp., Michigan
  - Oregon Medical Research Center, PC, Portland, Oregon
  - DermResearch, Inc., Austin, Texas
  - J & S Studies, Inc., College Station, Texas
  - Dermatology Treatment & Research Center, PA, Dallas, Texas
  - The Education & Research Foundation, Inc, Lynchburg, Virginia